CLINICAL TRIAL: NCT04869644
Title: A Personalized Trial Pilot to Test Habit Formation Theory for Low Intensity Physical Exercise in Older Adults
Brief Title: A Trial of Habit Formation Theory for Exercise in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Karina Davidson, Senior Vice President, Research & Dean of Academic Affairs, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-1182; P30AG063786-01 (NIH)
Record Dates: First submitted 2021-04-18; First posted 2021-05-03 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Sedentary Behavior; Aging; Activity, Motor; Behavior, Health
Keywords: Habit Formation; Physical Activity; Behavior Change; Virtual; Personalized Trial; Personalized; Feasibility
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Health Behavior | interventions — Organizational Objectives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Behavioral Change Techniques to encourage Habit Formation (Experimental): Individuals will receive daily text messages with the goal of increasing daily walking by 2,000 more steps 5 days per week. Participants will be enrolled for a baseline period lasting 2 weeks where their average daily activity level will be assessed using a Fitbit device to generate an average daily step counts. Following completion of baseline, participants will be asked to generate a walking plan with the goal of walking an additional 2,000 steps above their baseline activity level on 5 days per week. This walking plan will include details about day of the week, time of day, and location of walking. Once participants have completed their walking plan, they will receive daily texts based on the 5 identified BCTs for the duration of the 10-week intervention. All BCTs will be delivered daily. The goal of the text messages will be to encourage habit formation for walking behavior.
  Interventions: Behavioral: Goal setting; Behavioral: Action Planning; Behavioral: Self-monitoring of behavior; Behavioral: Behavioral Practice/Rehearsal; Behavioral: Habit Formation

INTERVENTIONS:
Behavioral: Goal setting — Goal setting: set or agree on a goal defined in terms of behavior to be achieved.
Behavioral: Action Planning — Action planning: prompt detailed planning of performance of behavior (must include a setting [walking to the mailbox], frequency, duration, and intensity.
Behavioral: Self-monitoring of behavior — Self-Monitoring of behavior: establish a method for person to monitor and record their number of steps based on their Fitbit.
Behavioral: Behavioral Practice/Rehearsal — Behavioral rehearsal: prompt practice or rehearsal of walking one or more times in a context when the performance may not be necessary, in order to increase habit and skill.
Behavioral: Habit Formation — Prompt rehearsal & repetition of walking 2,000 steps or more in the same context repeatedly so that the context elicits the behavior.

SUMMARY:
This personalized trial will evaluate the effects of five behavioral change techniques (BCTs) described in Habit Formation Theory (Goal setting, Action Planning, Self-Monitoring, Behavioral Practice/Rehearsal and Habit Formation) delivered by text message to enhance low-intensity walking by 2,000 more steps per day/5 days per week in healthy Northwell employees aged 45-75 years old.

DETAILED DESCRIPTION:
This pilot study uses a virtual, single-arm, personalized design to evaluate the effects of the five behavioral change techniques (BCTs) described in Habit Formation Theory (Goal Setting, Action Planning, Self-Monitoring, Behavioral Practice/Rehearsal and Habit Formation) delivered by text message to enhance low-intensity walking by 2,000 more steps per day/5 days per week in healthy Northwell employees aged 45-75 years old. Up to sixty participants will complete a 12-week personalized trial of their walking behavior and assess all five behavioral change techniques described in habit formation theory. Prior to beginning the trial, participants will be sent a Fitbit® activity tracking watch that monitors number of steps per day. Participants will be instructed to wear the Fitbit device all day and night, even when they are sleeping. The single-arm, personalized trial will be comprised of a 2-week baseline/screening phase and a 10-week intervention phase. During the baseline phase, participant's baseline levels of physical activity (operationalized as average steps per day measured using the Fitbit device) and adherence to the trial protocol (operationalized as wearing the Fitbit device for a minimum of 10 hours per day and completing daily survey measure) will be assessed. Participants who are adherent to the study protocol, defined as adherence to Fitbit use and survey measures on 80% or more days during baseline, will proceed to the intervention phase. At the beginning of the intervention, participants will develop a walking plan with the goal of walking 2,000 more steps per day than their average levels of baseline activity (e.g., if you walked an average of 6,000 steps per day during baseline, the new goal would be 8,000). The walking plan will include details about the day, time, and location of walking behavior. Participants will commit to walking according to this plan 5 days per week (e.g., walking 8,000 steps per day on 5 planned days. A time-sensitive text of all 5 BCTs will delivered to the participant when the context (e.g., day of week, time of day) that they pre-selected is encountered. Participants will later receive a text message with a link to a secure survey in which they will note whether they engaged with the five behavioral change techniques which were prompted. The goal of the intervention is to help participants make their walking behavior habitual and automatic. Participants will be assessed in terms of their satisfaction with the personalized trial design, their Fitbit-measured daily steps, adherence to their walking plan, and the automaticity of their walking behavior. After completion of the intervention phase, participants will be allowed to keep the Fitbit device.

ELIGIBILITY:
Inclusion Criteria:

Men and women who:

* Age 45 - 75 years old of age
* Fluent in English
* Employed in the Northwell Health system
* Community-dwelling
* Report they are in good general health, walk regularly and have never been informed by a clinician that it was not advisable/safe to participate in a low-intensity walking program
* Owns and can regularly access a smartphone capable of receiving text messages
* Owns and can regularly access an e-mail account

Exclusion Criteria for Factors that May Limit Adherence to Interventions or Affect Conduct of the Trial

* < 45 years old or > 75 years old
* Unable to speak/comprehend English
* Not employed in Northwell Health system
* Have self-reported poor health, limited mobility and/or have been advised by a clinician not to increase their low-intensity walking
* Pregnancy
* Previous diagnosis of a serious mental health condition or psychiatric disorder, such as bipolar disorder

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina W Davidson, Principal Investigator — Northwell Health
Locations (1):
- Center for Personalized Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including he statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to beginning the intervention, participants completed a 2-week baseline period. Data were collected for the overall BCT intervention, not for individual BCT messages. All BCTs were delivered simultaneously as a multi-BCT package.
Groups:
- Intervention: Behavioral Change Techniques to Encourage Habit Formation: Participants in Group 1 received BCT messages 5 days a week for a 10-week intervention period with the following BCTs: goal setting, action planning, self-monitoring of behavior, behavioral rehearsal, rehearsal conducted in a consistent context
Period: Assessed for Eligibility
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Started | 114
Did Not Meet or Complete Inclusion Criteria | 35
Did Not Consent to Study | 30
Completed | 49
Not Completed | 65
Period: Enrolled in Study
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Started | 49
Withdrew From Study | 5
Completed | 44
Not Completed | 5
Period: Baseline
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Started | 44
Ineligible After Baseline | 8
Withdrew From Study | 2
Completed | 34
Not Completed | 10
Period: Intervention
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Started | 34
Discontinued Intervention | 2
Completed | 32
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Of those enrolled in the study, 44 participants began baseline assessment.
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Number analyzed (Participants) | 44
Age, Customized [Count of Participants; unit: Participants]
  45 to 55 | 12
  46 to 65 | 26
  66 to 75 | 6
  Over 75 | 0
  Declined to Respond | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 1
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Automaticity Score.
Description: Automaticity of behavior is assessed by a 4-item questionnaire asking about the automaticity of participant's walking behavior using a 4-point Likert scale with responses ranging from "Strongly Disagree" to "Strongly Agree". Items are summed together to form a total score ranging from 0 to 12, with higher scores indicating that participant's new walking behaviors have become more habitual and automatic. Change in daily automaticity levels over the course of the intervention period will be examined until scores level out and reach a score of 8 or more on 7 consecutive days. Participants will be judged to have reached an asymptote at this point in time. The proportion of the sample that has achieved automaticity will be reported as a number with percentage [N(%)]. Time-to-event analyses will be conducting examining participant differences in reaching an asymptote for automaticity and overall time-to-event will represented using Kaplan-Meier curves.
Time Frame: Assessed daily via online survey for participants across the duration of the 10-week intervention. Daily assessments will be aggregated by week to generate weekly means for automaticity.
Population: Participants who completed the baseline eligibility period continued on to the intervention. All participants in the intervention period received the daily automaticity survey for the 10-week intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Number analyzed (Participants) | 34
Participants | 17

2. Primary Outcome: Participant Satisfaction With Personalized Trial Components.
Description: Participants will rate their satisfaction with the Personalized Trial overall and with individual elements of the trial in a satisfaction survey developed for this trial. Participants will rate 9 items assessing satisfaction with methods and process of the trial on a 4-point Likert scale with responses ranging from "0 - Not at all satisfied" to "3 - Very satisfied". Higher scores indicate greater levels of satisfaction. Means and standard deviations will be reported for each element of satisfaction.
Time Frame: Assessed once after completion of the study at 12 weeks.
Measure: Mean (Standard Deviation); unit: Score for Participant Satisfaction Item
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
Number analyzed (Participants) | 32
Score for Participant Satisfaction Item
  "Please rate your overall satisfaction with the BCT text messages" | 2.53 (0.78)
  "Please rate your satisfaction with the ease of using the BCT text messages" | 2.97 (0.18)
  "Please rate your satisfaction with the overall effectiveness of the BCT text messages" | 2.50 (0.82)
  "Video explanations and demonstrations of study devices and procedures" | 2.38 (0.67)
  "Text messaging for reminders (e.g. synch your Fitbit)" | 2.76 (0.54)
  "Text messaging for data collection (i.e. surveys)" | 2.65 (0.67)
  "Use of the Fitbit device to track your activity and sleep" | 2.60 (0.60)
  "Study communications" | 2.67 (0.58)
  "Presentation of your results" | 2.38 (0.92)

3. Secondary Outcome: Within-person Change in Daily Steps.
Description: Participant steps will be assessed continuously using a Fitbit mobile device. Daily steps for participants will be aggregated by baseline and intervention phases to generate average daily steps in each phase. Changes in daily steps between baseline and intervention phases will be compared using Generalized Linear Mixed Model analyses.
Time Frame: Steps will be assessed continuously via worn activity tracker and step counts will be reported daily.
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Days Adhering to Walking Habit.
Description: This is assessed using a single yes/no item assessed daily asking participants "Did you walk according to your walking plan today?". For each participant, we will identify the proportion of days during the 10-week intervention where the participant adhered to the walking plan. Proportions of adherence will reported across all participants with means and standard deviations.
Time Frame: Assessed once after completion of the study at 12 weeks.
Reporting Status: Not Posted

5. Secondary Outcome: Participant Attitudes and Opinions Towards Personalized Trials.
Description: Participants will be asked via survey about their attitudes and opinions regarding the personalized trial implementation (e.g., Did the trial feel burdensome?). Participants will rate items on a 7-point Likert scale with responses ranging from "0 - Strongly Disagree" to "6 - Strongly Agree". Higher scores indicate greater levels of agreement. Scores on each item will be reported with means and standard deviations.
Time Frame: Assessed once after the completion of the intervention period.
Reporting Status: Not Posted

6. Secondary Outcome: Participant Adherence to Self-Monitoring.
Description: This will be measured via a single survey item delivered following a participant's scheduled walking time asking them to record the number of steps they took on their walk. Individuals who complete this item and record their steps will be judged to be adherent to self-monitoring of their walking behavior. Participant adherence will be aggregated over the course of the 10-week intervention and will be reported as proportion of days adherent to self-monitoring. Proportions of adherence will be reported across all participants with means and standard deviations.
Time Frame: Assessed daily via online survey for participants across the duration of the 10 week intervention. Daily responses will be aggregated across the intervention to determine an overall proportion of days adherent self-monitoring of behavior.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data for adverse events were collected for each participant over 12 weeks (2-week baseline and 10-week intervention).
Arm/Group | Intervention: Behavioral Change Techniques to Encourage Habit Formation
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 2/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Behavioral Change Techniques to Encourage Habit Formation (N=44)
Rash (Product Issues) | 2 (2) — Participant developed a rash from wearing the Fitbit device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04869644/Prot_SAP_000.pdf